CLINICAL TRIAL: NCT00771199
Title: An Open-label, Multicenter Study to Evaluate the Safety/Tolerability and Clinical Utility of Low-dose TTS-Fentanyl D-TRANS in Taiwan Patients With Cancer Pain
Brief Title: An Efficacy and Safety Study of Low-dose Transdermal Therapeutic System (TTS)-Fentanyl D-Trans in Taiwan Participants With Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014602; FENPAI4054 (Other: Janssen-Cilag Ltd)
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Cancer, Pain
Keywords: Cancer pain; Pain; Fentanyl; Durogesic; Cancer; Transdermal
MeSH Terms: conditions — Cancer Pain; Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Therapeutic System (TTS)-Fentanyl (Experimental)
  Interventions: Drug: Transdermal Therapeutic System (TTS)-Fentanyl

INTERVENTIONS:
Drug: Transdermal Therapeutic System (TTS)-Fentanyl — Participants will receive 1 transdermal patch of TTS-fentanyl containing 12 micrograms per hour (mcg/h) for 28 days. Dose can be increased or decreased as per Investigator's discretion up to 100 mcg/h.

SUMMARY:
The purpose of this study is to evaluate safety/tolerability and clinical utility of low-dose transdermal therapeutic system (TTS [medicated adhesive pad that is placed on the skin to deliver a timed-release dose of medication through the skin into the bloodstream]) - fentanyl in Taiwan participants with cancer pain. Secondly, to demonstrate the dropout rate that will be decreased by initiating therapy with12 microgram per hour (mcg/hr) instead of with 25 mcg/h.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (when more than one hospital or medical school team work on a medical research study), single-arm, non-randomized study to evaluate the efficacy and safety of low-dose TTS-fentanyl in Taiwan participants with cancer pain. Eligible participants will be enrolled and scheduled to return at Day 0, 7, 14 and 28. Participants will receive TTS-fentanyl for 28 days at a starting dose of 12 micrograms per hour (mcg/h) (one patch). Dose of fentanyl can increased or decreased as per Investigator's discretion to maintain participant's pain score at 2 or less on the Brief Pain Inventory (BPI) question 6 (that tells how much pain you have right now). Safety will primarily be evaluated by measuring participant's dropout rate due to adverse events. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with cancer; histologically (examination of tissue specimens under a microscope) confirmed malignancy (term for diseases in which abnormal cells divide without control and can invade nearby tissues)
* Participants who are able to communicate effectively with study personnel
* Participants who have intolerable cancer pain (pain score greater than or equal to [>=] 4)
* Participants who have an estimated life expectancy of at least 30 days
* Participants who have given written dated informed consent to participate in the study

Exclusion Criteria:

* Participants who have already received regular treatment with an strong opioid (morphine-like synthetic narcotic that produces the same effects as drugs derived from the opium poppy [opiates]), for their pain before entering the study
* Participants who have already received tramadol (a narcotic-like pain reliever used to treat moderate to severe pain) treatment over 200 milligram (mg) for their pain before entering the study
* Participants with significant abnormalities in hepatic or renal function which would, in the opinion of the Investigator, prevent the participants involvement in the study
* Participants with significant clinical abnormalities in central nervous system (CNS), respiratory or cardiovascular function, which in the investigators judgment prevents participation in the study
* Pregnant or lactating females or females of child bearing potential not currently practicing documented, adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Dropped From Study due to Adverse Events | Day 0 up to Day 28
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical product. An adverse event does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. Percentage of participants who will be prematurely withdrawn from the study due to any adverse events will be reported.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) Score (Question 6) | Day 0, Day 7, Day 14 and Day 28
  The BPI question number 6 describes pain severity, will be measured by the daily pain diary on numeric rating scale (NRS), ranging from 1 to 10; where 0 signifies no pain and 10 signifies extreme pain.
BPI Score (Question 9) - Quality of Life (QOL) | Day 0, Day 7, Day 14 and Day 28
  Participant's quality of life (QOL) will be assessed by BPI question number 9 (items 9a to 9g), which describes "how during the past 24 hours pain has interfered with participants general activity, mood, walking ability, normal work, relation with other people, sleep, enjoyment of life". Each item will be measured on NRS, ranges from 1 to 10 where 0 signifies does not interfere and 10 signifies completely interferes. Total score is the average of scores of all items and ranges from 0 to 10, where higher scores signifies higher pain/interference.
Average Daily Dose and Final Dose of Transdermal Therapeutic System (TTS)-fentanyl | Day 0 up to Day 28
  The TTS-fentanyl dosage is only increased in consultation with the treating physician and according to the participant's analgesic requirements, with the intention of maintaining his/ her pain score at 2 or less on the BPI question 6.
Investigator's Global Assessment Scale Score | Day 0 and Day 28
  Investigator will complete a global assessment of the participants treatment with respect to pain control using 4-point scale, where 1 signifies poor, 2 signifies fair, 3 signifies good, 4 signifies very good.
Percentage of Participants With Treatment Satisfaction | Day 0 and Day 28
  Participants will rate their assessment of treatment satisfaction, using 4-point scale where 1 signifies poor, 2 signifies fair, 3 signifies good and 4 signifies very good.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.